CLINICAL TRIAL: NCT04001790
Title: Effect of a 9-Month Internship Intervention for Military Dependents With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20008778; CDMRP AR150172 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-06-20; First posted 2019-06-28 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Transition to Employment; Employment; Project Search Plus ASD Supports
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This is a randomized, wait-list controlled study of the efficacy of the Project Search plus ASD Supports Model (PS-ASD) in 32 adolescents and young adults aged 18 to 21 with autism spectrum disorder. Approximately 32 subjects will be enrolled and randomized in a 1:1 ratio to treatment or wait-list control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Search + ASD Supports (Experimental): Project SEARCH is an intensive 9-month job training program where youth with developmental disabilities in their last year of high school are embedded in a large community business such as a hospital, government complex, or banking center where they rotate through three 10-12 week internships within the business learning marketable skills, social communication, and adaptive behavior in the business setting. In order to meet the unique needs of youth with ASD, Wehman, et al. (2014) enhanced the Project SEARCH model by adding autism supports to the original model. Those added supports were: 1) on-site, intensive, systematic instruction using the principles of applied behavior analysis, 2) on-site support and consultation from a behavior/autism specialist, and 3) intensive staff training in ASD and the Project SEARCH Model.
  Interventions: Behavioral: Project Search plus ASD Supports
- Business as Usual (No Intervention): Business as Usual means these youth remain in their high school programs as determined on their individualized education plans

INTERVENTIONS:
Behavioral: Project Search plus ASD Supports — Nine month job training program embedded on Fort Eustis military base.
  Other Names: PS+ASD
  Arms: Project Search + ASD Supports

SUMMARY:
The aims of the project are: 1. VCU will modify the Project SEARCH Plus ASD Model to meet the needs of military dependents with ASD. 2. VCU will implement the intervention based upon the Project SEARCH plus ASD Supports manual and will measure fidelity of implementation. 3. VCU will measure the impact of the intervention on the social communication, behavioral adjustment and employment outcomes of the military dependents who participate compared to an equal control group who do not receive the intervention. Aim 1 is accomplished, and Aims 2 and 3 have been implemented. The Project SEARCH program is currently in its second year at the 773rd Mission Support Group, Joint Base Langley Eustis, Fort Eustis site. Additionally, all recruitment activities were completed for the second cohort of the project, with a total of 14 treatment group participants and 21 control group participants across the two cohorts thus far. In addition, all collaborating agencies have signed the memorandum of understanding. The relocation and deployment plan is currently is being piloted.

DETAILED DESCRIPTION:
Background: Young people with ASD present unique challenges related to post school employment outcomes. Competitive employment rates for individuals with ASD, regardless of intellectual ability, reportedly range between 4.1 to 11.8%. Across the ability spectrum, individuals with ASD have lower rates of participation in vocational or technical education, employment, and post-secondary education in 2 or 4-year programs than their peers with other disabilities. The findings from this literature indicate individuals with ASD continue to have significant challenges in all environments related to social interaction and communication into adolescence and adulthood. Military offspring present a particular risk for poor outcomes due to the mobile nature of their parents' jobs. This greatly impacts the individual with ASD who may not be able to access programs to assist them in the transition to employment as well as their parents who may not be able to take advantage of promotions that involve moving.

Objective/Hypothesis: The objective of this proposed project is to study the impact of Project SEARCH plus ASD Supports (PS-ASD) on the social communication, behavioral, and employment outcomes of military dependents with ASD across three vocational domains (employment status, wage, number of hours worked per week) and three personal domains (social responsiveness, mental health, and quality of life).

The six hypotheses driving this project propose that Young adults who participate in an employer-based employment training and placement program will: demonstrate a higher rate of employment, work more hours, and earn a higher wage than those in the control condition. Additionally, young adults who participate in a work-based employment training and placement program will increase their social responsiveness, display lower anxiety and depression scores, and report higher quality of life scores than those in the control condition.

Specific Aims: Aim 1. VCU will modify the Project SEARCH Plus ASD Model to meet the needs of military dependents with ASD.

Aim 2. VCU will implement the intervention based upon the Project SEARCH plus ASD Supports manual and will measure fidelity of implementation.

Aim 3. VCU will measure the impact of the intervention on the social communication, behavioral adjustment and employment outcomes of the military dependents who participate compared to an equal control group who do not receive the intervention.

Study Design: This is a randomized, wait-list controlled study of the efficacy of the Project Search plus ASD Supports Model (PS-ASD) in 32 adolescents and young adults aged 18 to 21 with autism spectrum disorder. Approximately 32 subjects will be enrolled and randomized in a 1:1 ratio to treatment or wait-list control groups. A sufficient number of potential subjects will be screened to achieve this number of enrolled subjects.

Clinical Impact: The PS-ASD model provides an option for youth with ASD who seek employment upon graduation from high school by providing high numbers of trials of vocational, social communication, and self-management skills using applied behavior analysis in the settings where those skills will be used. Immersion in a 9-month internship program via PS+ASD appears to improve self-management, independence, social responsiveness, work skills, and quality of life but further research like the proposed project is required to observe the impact of this model for military dependents with ASD. This proposed project will assist professionals and military personnel in identifying viable treatment models for military dependents in transition to adulthood. This is a critical need for this population of youth who frequently do not receive such intensive transition services.

ELIGIBILITY:
Inclusion Criteria:

* Has an ASD
* Between 18 - 21 years old
* Seeking community based employment upon graduation from high school
* Attends participating school
* Eligible for funding through the Virginia Department of Aging and Vocational Rehabilitation
* Has personal independence
* Is able to pass a drug screen and felony record check and immunizations up-to-date for employment purposes
* Is military dependent or connected

Exclusion Criteria:

* Unable to provide consent or assent
* Does not meet inclusion criteria

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wehman, PhD, Principal Investigator — Virginia Commonwealth University; Carol M Schall, PhD, Study Director — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
VCU will share de-identified data with the National Database for Autism Research (NDAR) after reviewing and receiving informed consent with participants. VCU will only share data if participants consent. VCU will not share any data that will reveal participant identity. VCU will assign a random number to all data that is different than any other number or code associated with data shared. Participants can refuse permission to share their data and continue to be in the study. Participants can also change their mind about sharing data at any point until the investigators close the study with our VCU Institutional Review Board.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: End of the study and will be available indefinitely
Access Criteria: Researchers with access to the NDAR database
URL: http://nda.nih.gov/

REFERENCES:
- [Result] Whittenburg HN, Schall CM, Wehman P, McDonough J, DuBois T. Helping High School-Aged Military Dependents With Autism Gain Employment Through Project SEARCH + ASD Supports. Mil Med. 2020 Jan 7;185(Suppl 1):663-668. doi: 10.1093/milmed/usz224. PMID 31498390
- See also: website describing project — http://vcurrtc.org/deployed2work/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Project Search + ASD Supports | Business as Usual
Started | 22 | 26
Completed | 21 | 24
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Project Search + ASD Supports | Business as Usual | Total
Number analyzed (Participants) | 22 | 26 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 26 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 18 | 23 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 11 | 15 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Competitive Integrated Employment Rates
Description: Increase in number of participants engaged in Full or part time work for minimum wage or higher with the same wages and benefits accorded to non-disabled workers in the same position and fully integrated with co-workers and customers without disabilities.accorded to non-disabled workers in the same position and fully integrated with co-workers and customers without disabilities.
Time Frame: baseline to 18 months
Population: Employed at 18 months
Measure: Count of Participants; unit: Participants
Groups:
- Project Search + ASD Supports: Project SEARCH is an intensive 9-month job training program where youth with developmental disabilities in their last year of high school are embedded in a large community business such as a hospital, government complex, or banking center where they rotate through three 10-12 week internships within the business learning marketable skills, social communication, and adaptive behavior in the business setting. In order to meet the unique needs of youth with ASD the study team enhanced the Project SEARCH model by adding autism supports to the original model. Those added supports were: 1) on-site, intensive, systematic instruction using the principles of applied behavior analysis, 2) on-site support and consultation from a behavior/autism specialist, and 3) intensive staff training in ASD and the Project SEARCH Model.
  Project Search plus ASD Supports: Nine month job training program embedded on Fort Eustis military base.
Arm/Group | Project Search + ASD Supports | Business as Usual
Number analyzed (Participants) | 20 | 18
Participants | 12 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Project Search + ASD Supports | Business as Usual
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/26
Other Adverse Events (participants affected / at risk) | 0/22 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04001790/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT04001790/ICF_000.pdf